CLINICAL TRIAL: NCT07335939
Title: Late-term Abortions Between 14 and 16 Weeks of Gestation: Comparison of Hemorrhagic Risks in Surgical vs. Medical Abortions
Acronym: IVG-Tardives
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9690
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Abortion Late
Keywords: Abortion Late; Ongoing single pregnancy; Ongoing multiple pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the extension of the legal abortion limit to 16 weeks by the law of March 2, 2022, we must adapt our care to reduce the risks associated with this procedure. According to the French National Authority for Health (HAS), all abortions after 9 weeks of gestation should be performed surgically, but the French National College of Gynecologists and Obstetricians (CNGOF) indicates that each patient should have the choice of method regardless of the gestational age at the time of the abortion.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman
* Single or multiple pregnancy
* Undergoing an abortion between 14 and 16 weeks of gestation at the Strasbourg University Hospital between March 2, 2022, and March 2, 2026

Exclusion Criteria:

* Missed Pregnancy
* Term < 14 Weeks of Gestation or > 16 Weeks of Gestation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: - Adult woman with single or multiple pregnancy and undergoing an abortion between 14 and 16 weeks of gestation at the Strasbourg University Hospital between March 2, 2022, and March 2, 2026
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Bleeding (in cc) | During surgery
  Bleeding > 500 cc means a very large blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie-Obstétrique - CHU de Strasbourg - France, Strasbourg, France